CLINICAL TRIAL: NCT05935189
Title: Establishment of a Tissue Registry for Hepatocellular Carcinoma Specimens for Genetic and Histologic Research
Brief Title: Establishment of a Tissue Registry for Hepatocellular Carcinoma Specimens
Acronym: TIR-HCC
Status: Recruiting | Type: Observational
Sponsor: Nikomed Medical Center (Network)
Responsible Party: Sponsor
Other Study IDs: NMC-2301
Record Dates: First submitted 2023-06-20; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — i. Tumor and liver tissue samples resulting from surgical/biopsy resection ii. 10 mL of whole blood collected on EDTA iii. Stool samples for further gut microbiota profiling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the study is to establish a cancer registry to facilitate research and assist in the identification of additional risk factors for hepatocellular carcinoma. The main objectives are:

1. provide a mechanism to store the information about subjects with hepatocellular carcinoma
2. use of tissue samples for translational/further research purposes

DETAILED DESCRIPTION:
The Establishment of a Tissue Registry for Hepatocellular Carcinoma biopsy specimens for genetic and histologic research (TIR-HCC) is a project aimed at addressing the high incidence rates of primary liver cancer in Armenia. This initiative seeks to establish a cancer registry to support research efforts and identify additional risk factors associated with hepatocellular carcinoma (HCC).

The study will involve patients of Armenian descent who exhibit clinical, biochemical, and imaging evidence of hepatocellular carcinoma. Data collection will include tissue and blood samples, which will undergo histologic and genetic analyses. Additionally, relevant clinical history, laboratory results, imaging findings, and gut microbiota profiles will be collected.

To ensure a comprehensive dataset, samples will be collected from eight institutions in Armenia. The project aims to accumulate data from a total of 500 patients, providing a substantial pool for research and analysis.

By establishing the TIR-HCC registry, researchers hope to contribute to the understanding of hepatocellular carcinoma and potentially identify new risk factors associated with the disease. The collected data will aid in advancing knowledge of HCC and guide future strategies for prevention, early detection, and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-confirmed diagnosis of HCC
* Armenian descent
* Having given their signed Informed consent

Exclusion Criteria:

* Failure to obtain informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is composed of individuals from Armenian descent who have a biopsy-confirmed diagnosis of hepatocellular carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Creation of a registry | 5 year
  The primary outcome of this study is to provide a mechanism to store the information about subjects with hepatocellular carcinoma. The outcome will be measured by the number of patients involved in the registry, measured by absolute numbers. The target number is 500 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hasmik Ghazinian, MD, Principal Investigator — Nikomed Medical Center
Locations (1):
- Nikomed Medical Center, Yerevan, Armenia

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- See also: Sung H, Ferlay J, Siegel RL, et al. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021;71(3):209-249. doi:10.3322/caac.21660 — https://pubmed.ncbi.nlm.nih.gov/33538338/

DOCUMENTS (1):
  • Study Protocol (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT05935189/Prot_000.pdf